CLINICAL TRIAL: NCT07138625
Title: Nebulized 3% Hypertonic Saline Versus Normal Saline in Managing Children With Acute Bronchiolitis: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Anbar (Other)
Responsible Party: Principal Investigator, Raid M. Al-Ani, Professor, University Of Anbar
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRC-1
Record Dates: First submitted 2025-08-16; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Bronchiolitis
Keywords: Nebulized 3% hypertonic saline; Nebulized normal saline; Acute bronchiolitis; Children; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nebulized 3% hypertonic saline (Active Comparator): Nebulized normal saline
  Interventions: Biological: Nebulized normal saline

INTERVENTIONS:
Biological: Nebulized normal saline — Eligible patients with moderate bronchiolitis who met the inclusion criteria were randomly assigned in a 1:1 ratio to either the hypertonic saline (3%) group or the normal saline (0.9%) group. Randomization was performed using a computer-generated random number sequence prepared by an independent statistician not involved in patient recruitment or treatment. Allocation concealment was ensured through the use of sequentially numbered, opaque, sealed envelopes, which were opened only after patient enrollment and completion of baseline assessments.

SUMMARY:
This randomized controlled trial was conducted at A-Ramadi Teaching Hospital for Maternity and Children on patients admitted with acute bronchiolitis. The study covered a duration of 6 months. The study was approved by the Ethical Approval Committee of the University of Anbar. Informed consent was obtained from each parent.

The severity of bronchiolitis was assessed based on the absence (score = 0) or presence (score = 1) of the following parameters: tachycardia, wheezing, use of accessory muscles, low oxygen saturation (SpO₂ < 95%), and feeding difficulties. The total score, therefore, ranged from 0 to 5. Severity was subsequently classified into three categories: Mild (0-1), patients typically discharged home without the need for hospitalization; Moderate (2-3), patients admitted to the general pediatric ward for closer observation and supportive care; and Severe (4-5), patients requiring admission to the PICU due to significant respiratory compromise, such as oxygen saturation < 90%, intercostal recession, and wheezing requiring respiratory support [15].

All patients aged 0-24 months with a clinical diagnosis of bronchiolitis, defined by signs of acute respiratory distress, chest radiographic findings consistent with bronchiolitis, and a bronchiolitis severity score of (2-3), whose parents or guardians provided informed consent were enrolled in the study. Exclusion criteria were: severely ill infants requiring mechanical ventilation; age greater than 2 years; presence of chronic illnesses such as chronic renal disease, congenital heart disease, or neuromuscular disorders; immunocompromised status (including malnutrition or chronic corticosteroid use); diagnosis of asthma; prior use of corticosteroids or bronchodilators; and refusal of caregivers to participate in the trial.

We calculate the required sample size according to the mean LOS of 3 days from a previous study [5] and aimed to detect a clinically meaningful 25% reduction (~0.75 days), with a standard deviation of 1.92 days, 90% power, and a two-sided alpha of 0.05. Using the two-sample t-test formula for comparing means, this resulted in approximately 139 patients per group, which was increased to 150 per group to account for potential dropouts.

Eligible patients with moderate bronchiolitis who met the inclusion criteria were randomly assigned in a 1:1 ratio to either the hypertonic saline (3%) group or the normal saline (0.9%) group. Randomization was performed using a computer-generated random number sequence prepared by an independent statistician not involved in patient recruitment or treatment. Allocation concealment was ensured through the use of sequentially numbered, opaque, sealed envelopes, which were opened only after patient enrollment and completion of baseline assessments.

Due to the physical characteristics of the solutions, blinding of the nursing staff administering the nebulization was not feasible. However, the physicians responsible for clinical assessment and outcome evaluation were blinded to the treatment allocation to minimize observer bias. Parents or guardians were not informed of the specific solution used, and both groups received nebulization with an identical-appearing setup to maintain partial blinding at the patient and caregiver level.

Patients with moderate bronchiolitis were randomly allocated into two groups. The first group received 3% hypertonic saline as a diluent with salbutamol, whereas the second group received 0.9% normal saline as a diluent with salbutamol. Nebulization was administered via a compressed air-driven jet nebulizer four times daily by well-trained nursing staff under the supervision of on-call physicians. All other aspects of bronchiolitis management were provided similarly to both groups, including oxygen supplementation to maintain SpO₂ > 92%, airway suctioning, nebulization with salbutamol, and corticosteroid therapy. A follow-up flow chart was maintained for direct monitoring of each patient's clinical symptoms and signs of respiratory distress. Baseline clinical symptoms, vital signs, and respiratory severity scores were recorded for all participants at admission before initiation of the treatment protocol.

Data were analyzed using the Statistical Package for the Social Sciences software, version 29. Continuous variables were tested for normality using the Shapiro-Wilk test. Normally distributed data were expressed as mean±SD and compared between groups using the independent samples t-test. Non-normally distributed variables were presented as median and analyzed using the Mann-Whitney U test. Categorical variables were presented as frequencies and percentages, and differences between groups were assessed using the chi-square test or Fisher's exact test, as appropriate. The primary outcome was the difference in LOS between the two groups. Secondary outcomes included changes in respiratory severity score, oxygen saturation, and the proportion of patients progressing to severe disease.

DETAILED DESCRIPTION:
Introduction Bronchiolitis is an acute viral infection of the lower respiratory tract, most commonly caused by the respiratory syncytial virus (RSV). By the age of one year, more than 60% of children have been infected with RSV, and by the age of two years, the infection rate exceeds 90% [1].

Acute bronchiolitis typically occurs in epidemic outbreaks during the winter months. Pathologically, it is characterized by acute inflammation, edema, and necrosis of the epithelial lining of the bronchioles. These changes lead to excessive mucus production, which obstructs airflow and results in progressive deterioration of respiratory function [2].

Clinical presentation in bronchiolitis varies, it may present as enormous cough, rapid breathing, fever, acute wheeze or signs of respiratory compromise [3].

There are different risk factors leading to increased risk of severe bronchiolitis or hospitalization such as younger age infant, prematurity, congenital abnormality such as Downs syndrome, congenital heart disease, immunodeficiency, and chronic kidney disease [4].

In children with bronchiolitis, the median length of hospital stay (LOS) is approximately 3 days; however, admission to the pediatric intensive care unit (PICU) may be required in up to 5.6% of hospitalized cases. The mortality rate for bronchiolitis is estimated at 2.8 per 100,000 persons [5].

The severity of bronchiolitis is classified into three categories based on respiratory features and the need for intervention. Mild cases can be managed with supportive measures alone, while moderate and severe cases require hospitalization, oxygen therapy, and in some instances, mechanical ventilation via endotracheal intubation, along with supportive measures such as adequate hydration. Although treatment options such as corticosteroids and bronchodilators have been explored, their effectiveness in altering the disease course remains controversial [6].

Recently, several studies have focused on the benefits of hypertonic saline (3%), which facilitates the movement of water molecules into the lung mucosa, promotes their absorption by the bronchial and submucosal layers, and helps reduce the risk of airway edema formation [7-9]. By utilizing the principle of vaporization, hypertonic saline also helps moisturize the airway surface, enhance mucociliary function, and facilitate the clearance of obstructive sputum, thereby improving treatment outcomes [10].

Although many previous investigations, including systematic reviews and meta-analyses, have reported that hypertonic saline (3%) may reduce LOS and disease severity compared with normal saline, the findings remain inconsistent [11, 12]. Conversely, some studies have found no significant benefit of hypertonic saline (3%) over normal saline in children with acute bronchiolitis [13], whereas other investigations have demonstrated that hypertonic saline (3%) can reduce modified respiratory assessment scores and LOS [14]. Moreover, a recent systematic review and meta-analysis concluded that previous clinical trials on the management of acute bronchiolitis often excluded high-risk groups of children [4].

Owing to the severe shortage, and at times complete unavailability, of hypertonic saline (3%) in our hospital, most pediatricians routinely use nebulized normal saline as part of the standard management regimen for acute bronchiolitis. Therefore, this study was undertaken to evaluate the effect of nebulized 3% hypertonic saline compared with normal saline in hospitalized children with acute bronchiolitis, with particular focus on its impact on disease severity and LOS.

Material and method This randomized controlled trial was conducted at A-Ramadi Teaching Hospital for Maternity and Children on patients admitted with acute bronchiolitis. The study covered a duration of 6 months (October 2025-March 2026). The study was approved by the Ethical Approval Committee of the University of Anbar. Informed consent was obtained from each parent.

The severity of bronchiolitis was assessed based on the absence (score = 0) or presence (score = 1) of the following parameters: tachycardia, wheezing, use of accessory muscles, low oxygen saturation (SpO₂ < 95%), and feeding difficulties. The total score, therefore, ranged from 0 to 5. Severity was subsequently classified into three categories: Mild (0-1), patients typically discharged home without the need for hospitalization; Moderate (2-3), patients admitted to the general pediatric ward for closer observation and supportive care; and Severe (4-5), patients requiring admission to the PICU due to significant respiratory compromise, such as oxygen saturation < 90%, intercostal recession, and wheezing requiring respiratory support [15].

All patients aged 0-24 months with a clinical diagnosis of bronchiolitis, defined by signs of acute respiratory distress, chest radiographic findings consistent with bronchiolitis, and a bronchiolitis severity score of (2-3), whose parents or guardians provided informed consent were enrolled in the study. Exclusion criteria were: severely ill infants requiring mechanical ventilation; age greater than 2 years; presence of chronic illnesses such as chronic renal disease, congenital heart disease, or neuromuscular disorders; immunocompromised status (including malnutrition or chronic corticosteroid use); diagnosis of asthma; prior use of corticosteroids or bronchodilators; and refusal of caregivers to participate in the trial.

We calculate the required sample size according to the mean LOS of 3 days from a previous study [5] and aimed to detect a clinically meaningful 25% reduction (~0.75 days), with a standard deviation (SD) of 1.92 days, 90% power, and a two-sided alpha of 0.05. Using the two-sample t-test formula for comparing means, this resulted in approximately 139 patients per group, which was increased to 150 per group to account for potential dropouts.

Eligible patients with moderate bronchiolitis who met the inclusion criteria were randomly assigned in a 1:1 ratio to either the hypertonic saline (3%) group or the normal saline (0.9%) group. Randomization was performed using a computer-generated random number sequence prepared by an independent statistician not involved in patient recruitment or treatment. Allocation concealment was ensured through the use of sequentially numbered, opaque, sealed envelopes, which were opened only after patient enrollment and completion of baseline assessments.

Due to the physical characteristics of the solutions, blinding of the nursing staff administering the nebulization was not feasible. However, the physicians responsible for clinical assessment and outcome evaluation were blinded to the treatment allocation to minimize observer bias. Parents or guardians were not informed of the specific solution used, and both groups received nebulization with an identical-appearing setup to maintain partial blinding at the patient and caregiver level.

Patients with moderate bronchiolitis were randomly allocated into two groups. The first group received 3% hypertonic saline as a diluent with salbutamol, whereas the second group received 0.9% normal saline (isotonic) as a diluent with salbutamol. Nebulization was administered via a compressed air-driven jet nebulizer four times daily by well-trained nursing staff under the supervision of on-call physicians. All other aspects of bronchiolitis management were provided similarly to both groups, including oxygen supplementation to maintain SpO₂ > 92%, airway suctioning, nebulization with salbutamol, and corticosteroid therapy. A follow-up flow chart was maintained for direct monitoring of each patient's clinical symptoms and signs of respiratory distress. Baseline clinical symptoms, vital signs, and respiratory severity scores were recorded for all participants at admission before initiation of the treatment protocol.

Data were analyzed using the Statistical Package for the Social Sciences (SPSS) software, version 29 (IBM Corp., Armonk, NY, USA). Continuous variables were tested for normality using the Shapiro-Wilk test. Normally distributed data were expressed as mean ± SD and compared between groups using the independent samples t-test. Non-normally distributed variables were presented as median (interquartile range, IQR) and analyzed using the Mann-Whitney U test. Categorical variables were presented as frequencies and percentages, and differences between groups were assessed using the chi-square test or Fisher's exact test, as appropriate. The primary outcome was the difference in length of hospital stay (LOS) between the two groups. Secondary outcomes included changes in respiratory severity score, oxygen saturation, and the proportion of patients progressing to severe disease. For within-group comparisons over time, repeated measures analysis of variance (ANOVA) or the Friedman test (for non-parametric data) was applied. A P-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: All patients aged 0-24 months with a clinical diagnosis of bronchiolitis, defined by signs of acute respiratory distress, chest radiographic findings consistent with bronchiolitis, and a bronchiolitis severity score of (2-3), whose parents or guardians provided informed consent were enrolled in the study.

-

Exclusion Criteria: Exclusion criteria were: severely ill infants requiring mechanical ventilation; age greater than 2 years; presence of chronic illnesses such as chronic renal disease, congenital heart disease, or neuromuscular disorders; immunocompromised status (including malnutrition or chronic corticosteroid use); diagnosis of asthma; prior use of corticosteroids or bronchodilators; and refusal of caregivers to participate in the trial.

-

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the difference in length of hospital stay (LOS) between the two groups | 1-72 hours

IPD SHARING:
Plan to Share IPD: No